CLINICAL TRIAL: NCT05933499
Title: Effect of Tirzepatide and Bimagrumab on Body Composition, Insulin Sensitivity, and Bone in Adults With Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Melanie Schorr Haines, M.D, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P001334
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — bimagrumab; Tirzepatide; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomized in 1:1:1 ratio to tirzepatide 15mg SQ qweek + bimagrumab 300mg SQ qweek, tirzepatide 15mg SQ week, or bimagrumab 300mg SQ qweek,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide + bimagrumab (Experimental)
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide; Dietary Supplement: Calcium/Vitamin D; Behavioral: Lifestyle and nutrition counseling
- Tirzepatide + placebo (Active Comparator)
  Interventions: Drug: Tirzepatide; Dietary Supplement: Calcium/Vitamin D; Behavioral: Lifestyle and nutrition counseling
- Bimagrumab + placebo (Active Comparator)
  Interventions: Drug: Bimagrumab; Dietary Supplement: Calcium/Vitamin D; Behavioral: Lifestyle and nutrition counseling

INTERVENTIONS:
Drug: Bimagrumab — SQ bimagrumab 300mg qweek
  Arms: Bimagrumab + placebo; Tirzepatide + bimagrumab
Drug: Tirzepatide — SQ tirzepatide 15mg qweek
  Arms: Tirzepatide + bimagrumab; Tirzepatide + placebo
Dietary Supplement: Calcium/Vitamin D — Elemental calcium 1200 mg + vitamin D3 800 IU PO daily
Behavioral: Lifestyle and nutrition counseling — Lifestyle and nutrition counseling consistent with current guidelines for weight management

SUMMARY:
In adults with obesity seeking treatment, weight loss would ideally be composed almost exclusively of fat mass. However, loss of muscle mass and bone are unintentional consequences of weight loss, which may have negative effects on health by lessening improvements in glucose and insulin levels, reducing resting metabolic rate, and increasing the risk of falls and fractures. Data in animals and humans suggest that bimagrumab, an investigational new drug for obesity that inhibits the activin type II receptor (ActRII) inhibitor, may help maximize loss of fat mass while maintaining muscle mass when used in combination with a glucagon-like peptide 1 receptor agonist (GLP-1 RA). The investigators hypothesize that in a randomized, placebo-controlled trial of 63 adults with obesity randomized to tirzepatide (GLP-1/GIP RA) + bimagrumab, tirzepatide alone, or bimagrumab alone, the combination of tirzepatide + bimagrumab will result in improvements in muscle, fat, and bone compared to tirzepatide alone or bimagrumab alone when given in addition to a lifestyle intervention for weight loss over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2 or ≥27kg/m2 with at least one weight-related medical condition
* Have a history of at least one self-reported unsuccessful behavioral effort to lose body weight

Exclusion Criteria:

* Current or prior history of diabetes mellitus based on self-report, use of diabetes medications, HbA1c ≥6.5%, or fasting glucose ≥126 mg/dL
* Any single serum transaminase level (i.e., ALT, AST, alk phos) ≥3x the upper limit of normal (ULN)
* Serum lipase and/or amylase levels ≥2x ULN
* Serum bilirubin level >1.6 mg/dL
* Chronic kidney disease (e.g., estimated glomerular filtration rate (eGFR) < 45 mL/min)
* Total WBC <3000/μL, neutrophils <1500/μL, hemoglobin <12 g/dL, or platelet count <100,000/μL
* Significant coagulopathy, e.g., PT/INR >1.5
* History of familial hypertriglyceridemia or serum fasting triglyceride >500 mg/dL
* Uncontrolled thyroid disease, defined as abnormal TSH with abnormal fT4
* Any chronic active infection (e.g., HIV, hepatitis B or C) or hepatitis C treatment within the previous 6 months
* Known history or presence of severe active acute or chronic liver disease (e.g., cirrhosis) or conditions with hepatotoxic potential (e.g., gallbladder or bile duct disease, acute or chronic pancreatitis, exocrine pancreatic insufficiency)
* Active clinically significant gastric emptying abnormality or chronic use of a drug(s) that directly affect GI motility
* History of clinically significant arrhythmias, unstable angina, myocardial infarction, stroke, coronary artery bypass graft surgery, percutaneous coronary intervention, heart failure, valve disorders or defect, pulmonary hypertension, chronic hypotension (<100/50), or chronic uncontrolled hypertension (>160/100)
* Tachycardia, defined as heart rate >100 bpm after 5 minutes resting in a sitting position
* History of malignancy of any organ system (other than localized squamous or basal cell carcinoma of the skin), treated or untreated, within the previous 5 years
* Confirmed diagnosis of current, significant psychiatric disease (e.g., dementia, Alzheimer's disease, schizophrenia, or bipolar disorder). Individuals with adequately treated depression on stable treatment for at least 3 months are eligible.
* Prior history of suicide attempt
* PHQ-9 score ≥ 15 at screening
* Personal or family history of multiple endocrine neoplasia 2A or 2B or medullary thyroid cancer
* Active alcohol, drug, or tobacco abuse
* Have obesity induced by other endocrinologic disorders (e.g., Cushing syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., Melanocortin 4 Receptor deficiency or Prader Willi syndrome)
* History of weight loss surgery or planned weight loss surgery during the trial period
* Use of any anti-obesity medication, nutritional supplement, or over the counter (OTC) product for weight loss within the previous 6 months or during study participation
* Any new dietary intervention or exercise regimen for weight loss started within the previous 3 months
* Weight instability of >5kg within the previous 3 months
* Weight > 150kg due to limitations of radiology imaging machines
* Use of medications known or suspected to induce weight gain within the previous 3 months or during study participation (e.g., anti-androgens, gonadotropin releasing hormone (GnRH) analogs, some anticonvulsant and psychotropic medications (excluding anti-depressant medication) and oral glucocorticoids)
* Use of skeletal muscle anabolic agents within the previous 3 months or during study participation (e.g., hormones such as growth hormone or testosterone, nutritional supplements (other than protein) and over-the-counter products labeled as muscle anabolic agents)
* History of hypersensitivity to monoclonal antibodies or drugs in the same compound class as the study drugs
* Bone fracture within the previous 3 months
* Use of IV bisphosphonates within the previous 2 years or other osteoporosis medications within the previous 12 months or during study participation
* Not able or willing to comply with dietary and lifestyle intervention for weight loss, including history of clinically significant condition that precludes regular walking for exercise or contraindication to following a 500-calorie daily deficit, high protein diet
* Women who are pregnant or breastfeeding
* Women of child-bearing potential, defined as women physiologically capable of becoming pregnant, unless they are using an intrauterine device (IUD) from at least 3 months before the baseline visit through at least 4 months after the last drug dose and an additional contraceptive (barrier) method from screening through at least 4 months after the last drug dose. The following groups of women are eligible to participate: (a) women who are s/p surgical bilateral oophorectomy or total hysterectomy at least 6 weeks before taking study treatment, (b) women who have an IUD (see additional criteria above), (c) women who are s/p tubal ligation provided that they use an additional barrier form of contraception from screening through at least 4 months after the last drug dose, and (d) women who are post-menopausal defined as ≥12 months of spontaneous amenorrhea with appropriate clinical and hormonal profile (e.g., age-appropriate, history of vasomotor symptoms, and/or FSH >40 IU/L)
* For men, morning serum testosterone less than 200 ng/dL
* Concurrently enrolled in any other type of medical research judged to be scientifically or medically incompatible with this study
* Plans to move out of the study area within 16 months, or be out of the study area for >4 weeks, continuously
* Routine MRI exclusion
* Donation or loss of 400 mL or more of blood within past 2 months or plasma donation (> 250 mL) within past 2 weeks
* Any disorder, unwillingness, or inability not covered by any of the other exclusion criteria, which in the Investigator's opinion, might jeopardize the subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of kilograms of lean mass by dual-energy x-ray absorptiometry | 52 weeks
  Change in number of kilograms of lean mass by dual-energy x-ray absorptiometry in tirzepatide + bimagrumab vs. tirzepatide groups

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States